CLINICAL TRIAL: NCT01275352
Title: A Randomized, Double Blind Pilot Study Evaluating CLCNKA (Ka Renal Chloride Channel[ClC-Ka]) Polymorphism Effects on Hypertrophy Regression in Caucasian Hypertensive Patients Treated With Eplerenone
Brief Title: CLCNKA (Ka Renal Chloride Channel[ClC-Ka]) Polymorphism Effects on Hypertrophy Regression
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Thomas Cappola, MD, ScM, University of Pennsylvania
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLNCKA-1
Record Dates: First submitted 2011-01-10; First posted 2011-01-12 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Hypertension
Keywords: left ventricular hypertrophy; heart failure
MeSH Terms: conditions — Hypertension; Hypertrophy, Left Ventricular; Heart Failure | interventions — Eplerenone; Mineralocorticoid Receptor Antagonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (Active Comparator): Caucasian hypertensive patients who are homozygous for the ClC-Ka Gly/Gly83 allele
  Interventions: Drug: Eplerenone
- Arm 2 (Active Comparator): Caucasian hypertensive patients who are homozygous for ClC-Ka Arg/Arg 83 allele
  Interventions: Drug: Eplerenone
- Arm 3 (Placebo Comparator): Caucasian hypertensive patients who are homozygous for ClC-Ka Arg/Arg 83 allele
  Interventions: Drug: placebo
- Arm 4 (Placebo Comparator): Caucasian hypertensive patients who are homozygous for the ClC-Ka Gly/Gly83 allele
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Eplerenone — Eplerenone 50 mg/day
  Other Names: Inspra; aldosterone antagonist
  Arms: Arm 1; Arm 2
Drug: placebo — placebo
  Arms: Arm 3; Arm 4

SUMMARY:
This study will consist of middle-aged Caucasian non-failing subjects with high blood pressure who are homozygous for a gene that confers increased risk of developing heart failure, the Glycine 83 variant of the Ka renal chloride channel (ClC-Ka Gly/Gly 83), or middle-aged Caucasian non-failing hypertensive subjects who lack the heart failure risk gene, the wild-type Arginine 83 Ka renal chloride channel (ClC-Ka Arg/Arg 83). Subjects on standard therapy for high blood pressure with an angiotensin converting inhibitor (ACEI) or angiotensin receptor blocker (ARB) will be randomized to additional treatment with eplerenone (an aldosterone antagonist) or placebo, and assessed for changes in echocardiographic left ventricular hypertrophy (LVMI). Secondary endpoints will assess left ventricular remodeling and other echocardiographic variables. The investigators hypothesize that subjects homozygous for the CLCNKA risk allele will have a greater response to eplerenone in terms of reductions in LVMI than those lacking the risk allele.

DETAILED DESCRIPTION:
The screening phase will involve identifying Caucasian hypertensive patients who are homozygous for the ClC-Ka Gly/Gly83 and the ClC-Ka Arg/Arg 83 allele. All patients will be on background therapy with an angiotensin converting enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB) at least mid range dosing. If patient is not at recommended dose of ACE or ARB they must be titrated up and be stable on a midrange dose of ACEI or ARB for at least 4 weeks before they can be entered into the study. There will be 2 treatment phases. Phase 1 will be up to 4 weeks in duration and will consist of randomization to one table of eplerenone (25 mg) or matching placebo. On week 2 the patient will be up titrated to two tablets of eplerenone (50 mg) or matching placebo, to achieve a target dose of 50 mg of eplerenone. If the patient cannot tolerate two tablets of eplerenone or matching placebo they can be down titrated to one tablet of eplerenone or matching placebo. The target BP on study medication is < 130/80 mmHg. After the patients have been up titrated to the maximally tolerated dose of study medication, the background hypertension therapy can be adjusted to reach the target BP of < 130/80 mmHg by the end of week 4. Phase 2 will be 52 weeks in duration to assess the effects of placebo or eplerenone on LV hypertrophy. Serum potassium will be monitored throughout the study, and if necessary, doses of eplerenone will be titrated down as necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Caucasians with hypertension who are homozygous for the ClC-Ka Gly/Gly83 and the ClC-Ka Arg/Arg 83 allele.
2. Male or non-pregnant female aged 40 to 80 years.
3. Hypertension, defined as currently taking high blood pressure medications or not on medications but having SDP >140 or DBP >90.
4. Ejection fraction > 50% by any method within 6 months of the screening visit.
5. The Investigator must obtain written informed consent before the subject is screened for the study.
6. Subject should be on stable dose of ACE or ARB at moderate dosing for at least 4 weeks before randomization.

Exclusion Criteria:

1. History of heart failure with preserved or depressed ejection fraction.
2. Creatinine clearance of < 45 mL/min based on the Cockcroft-Gault formula (Appendix C).
3. Pregnancy
4. Life expectancy less than 12 months.
5. Planned cardiac surgery or percutaneous cardiac intervention within 3 months.
6. Serum potassium >5.5 mEq/L.
7. History of hyperkalemia (K>6.0 mEq/L) with eplerenone or spironolactone.
8. Myocardial infarction or stroke within 3 months of screening.
9. Evidence of clinical instability (hypotension, arrhythmias, unstable angina etc.).
10. Subjects on or requiring K-sparing diuretics or spironolactone.
11. Concomitant use of potent inhibitors of CYP3A4 including ketoconazole, itraconazole, nefazodone, troleandomycin, clarithromycin, ritonavir, and nelfinavir or any drug noted in the Contraindications, Warnings or Precautions sections of their labeling to be potent CYP3A4 inhibitors
12. Known hypersensitivity to eplerenone or spironolactone.
13. Evidence of current alcohol or drug abuse Severe organic disorders or surgery or disease of the gastrointestinal tract that in the opinion of the Investigator may interfere in the absorption and elimination of the study drug.
14. Psychoses or behavioral conditions that in the opinion of the Investigator would limit study compliance.
15. Subjects who have received any investigational medication or used any investigational device within 30 days prior to first dose of study drug or subjects actively participating in any investigational drug or device study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2014-12 (Estimated); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in LV mass index (g/m2) in ClC-Ka Gly/Gly83 patients and ClC-Ka Gly/Gly83 patients | 12 months

SECONDARY OUTCOMES:
Change in LV relative wall thickness | 6 and 12 months
Change in N-terminal pro-brain natriuretic peptide (NT-proBNP) | 6 and 12 months
Change in LV mass index (g/m2) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Cappola, MD, Principal Investigator — University of Pennsylvania; Gerald Dorn, MD, Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Barnes Jewish Hospital, St Louis, Missouri
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania